CLINICAL TRIAL: NCT04360447
Title: Comparison of the Effects of Reformer Pilates and Home Exercise Programs on Upper Extremity Muscle Strength in Paraplegic Patients: Prospective Randomized Controlled Study
Brief Title: Comparison of Pilates &Home Exercise Programs on Muscle Strength in Paraplegic Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IstPRMTRH
Record Dates: First submitted 2020-04-22; First posted 2020-04-24 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Spinal Cord Injuries
Keywords: spinal cord injuries; reformer pilates; home exercise
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Reformer pilates group (Experimental): Reformer pilates was planned, suitable for the disabled, with an instructor for the patients in the study group for 8 weeks.
  Interventions: Device: Reformer Pilates
- Home exercise group (Active Comparator): A home exercise program with telephone monitoring was planned for the patients in the control group for 8 weeks.
  Interventions: Other: Home Exercise

INTERVENTIONS:
Device: Reformer Pilates — Reformer pilates was planned, suitable for the disabled, with an instructor for the patients in the study group for 8 weeks.
  Arms: Reformer pilates group
Other: Home Exercise — A home exercise program with telephone monitoring was planned for the patients in the control group for 8 weeks.
  Arms: Home exercise group

SUMMARY:
Paraplegic patients to be included in the study were divided into 2 groups by randomization and it was planned to apply reformer pilates or home exercise programs for 8 weeks. It was aimed to compare upper extremity muscle strengths, Spinal Cord Independence Measure version III (SCIM-III) and the Short Form(36) Health Survey (SF-36) data before and after treatment.

DETAILED DESCRIPTION:
Spinal cord injuries (SCI) are injuries that occur as a result of compression, incision or contusion of the spinal cord, which extends from foramen magnum to cauda equina.These patients experience various complications and organ system damage in the chronic period.Their self-dependence is affected by the level of injury. One of the most important factors affecting the self-dependence of people with SCI is the strength of the upper extremity.Strong upper extremities are needed for independent transfer from bed.

SCI patients member of Turkish Spinal Cord Injury Association, according to the criteria for inclusion in the study patient list was created. In accordance with the sample size with the random numbers prepared with a computer program from this list, 18 people were planned to be included in the study. The patients were planned to be randomly divided into the study and control groups.Reformer pilates was planned, suitable for the disabled, with an instructor for the patients in the study group for 8 weeks; A home exercise program with telephone monitoring was planned for the patients in the control group for 8 weeks.It was planned to record the demographic data of the patients (age, gender, occupation, additional disease).It was planned to fill the SF-36 form to measure the quality of life of the patients, SCIM-III forms to evaluate functionally and measure the upper extremity muscle strength with a hand dynamometer.

At the end of 8 weeks, the patients were called for an examination, and SF-36, SCIM-III forms were filled and muscle strength was measured, and the comparison was aimed within the group and between the groups.In our study, our aim is to demonstrate the applicability of the reformer pilates program in SCI patients. In addition, to show the effects of home exercise program and reformer pilates programs on upper extremity muscle strength in SCI patients with multiple comparison tests.

ELIGIBILITY:
Inclusion Criteria:

* Volunteering for study
* Lesion level: T2 and below diagnosed with SCI
* Lesion duration over 2 years
* Ambulation in wheelchair
* To ensure randomization, SCI patients must be a member of Turkish Spinal Cord Injury Association and which should not be included in any study group.

Exclusion Criteria:

* Severe psychiatric disorder
* General condition disorder (heart failure, lung failure)
* Intolerably shoulder pain during exercise

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
the upper extremity muscle strength | 8 weeks
  measure the upper extremity muscle strength with a hand dynamometer

SECONDARY OUTCOMES:
the Short Form(36) Health Survey (SF-36) | 8 weeks
  The SF-36 is a measure of health status.It consists of eight scaled scores, which are the weighted sums of the questions in their section. The lower the score the more disability.
Spinal Cord Independence Measure version III (SCIM-III) | 8 weeks
  SCIM-III is a measurement tool for determining the level of function in spinal cord injury

CONTACTS AND LOCATIONS:
Overall Officials: Fatma N Kesiktaş, Assoc. Prof, Principal Investigator — Istanbul Physical Medicine Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine Rehabilitation Training and Research Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Dost G, Dulgeroglu D, Yildirim A, Ozgirgin N. The effects of upper extremity progressive resistance and endurance exercises in patients with spinal cord injury. J Back Musculoskelet Rehabil. 2014;27(4):419-26. doi: 10.3233/BMR-140462. PMID 24614829
- [Background] Yildirim A, Surucu GD, Karamercan A, Gedik DE, Atci N, Dulgeroglu D, Ozgirgin N. Short-term effects of upper extremity circuit resistance training on muscle strength and functional independence in patients with paraplegia. J Back Musculoskelet Rehabil. 2016 Nov 21;29(4):817-823. doi: 10.3233/BMR-160694. PMID 27002667
- [Background] Sipski ML, Richards JS. Spinal cord injury rehabilitation: state of the science. Am J Phys Med Rehabil. 2006 Apr;85(4):310-42. doi: 10.1097/01.phm.0000202105.87011.bf. No abstract available. PMID 16554684
- [Background] Kirshblum SC, Burns SP, Biering-Sorensen F, Donovan W, Graves DE, Jha A, Johansen M, Jones L, Krassioukov A, Mulcahey MJ, Schmidt-Read M, Waring W. International standards for neurological classification of spinal cord injury (revised 2011). J Spinal Cord Med. 2011 Nov;34(6):535-46. doi: 10.1179/204577211X13207446293695. No abstract available. PMID 22330108
- [Background] Gibson KL. Caring for a patient who lives with a spinal cord injury. Nursing. 2003 Jul;33(7):36-41; quiz 42. doi: 10.1097/00152193-200307000-00031. No abstract available. PMID 12851498
- [Background] Jacobs PL, Nash MS. Exercise recommendations for individuals with spinal cord injury. Sports Med. 2004;34(11):727-51. doi: 10.2165/00007256-200434110-00003. PMID 15456347